CLINICAL TRIAL: NCT06303414
Title: Revascularization for Symptomatic Non-acute Carotid Artery Occlusion
Acronym: RESCO
Status: Recruiting | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Other Study IDs: RESCO
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2016-06

CONDITIONS: Non-acute Carotid Artery Occlusion
MeSH Terms: interventions — Endarterectomy, Carotid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Carotid Endarterectomy (CEA): Patients who are treated with CEA.
  Interventions: Procedure: Carotid Endarterectomy (CEA)
- Carotid Artery Stenting (CAS): Patients who are treated with CAS.
  Interventions: Procedure: Carotid Artery Stenting (CAS)
- Hybrid Surgery: Patients who are treated with Hybrid Surgery.
  Interventions: Procedure: Hybrid Surgery

INTERVENTIONS:
Procedure: Carotid Endarterectomy (CEA) — Carotid endarterectomy (CEA) Surgeons follow the contemporary guideline combined with their experience and preference in order to ultimately select what is best suited for the patient and choose between CEA, CAS and Hybrid Sugery. Patients will receive 100 mg of aspirin or 75 mg of clopidogrel daily starting from at least 72 h prior to the CEA procedure and continued receiving the medication indefinitely. General anesthesia is recommended for CEA, although the use of standard or eversion endarterectomy, and a shunt or patch, is left to the discretion of the surgeon.
  Groups: Carotid Endarterectomy (CEA)
Procedure: Carotid Artery Stenting (CAS) — Carotid artery stenting (CAS) Surgeons follow the contemporary guideline combined with their experience and preference in order to ultimately select what is best suited for the patient and choose between CEA, CAS and Hybrid Sugery. Patients will be given 100 mg of aspirin plus 75 mg of clopidogrel daily for at least 3 days before the CAS procedure and for 90 days after the procedure. They will receive a daily dose of 100 mg aspirin or 75 mg clopidogrel thereafter. For the CAS procedure, general anesthesia and predilation prior to stent placement are recommended. Use of an embolic protection device is advised for all patients who undergo CAS.
  Groups: Carotid Artery Stenting (CAS)
Procedure: Hybrid Surgery — Hybrid Surgery Surgeons follow the contemporary guideline combined with their experience and preference in order to ultimately select what is best suited for the patient and choose between CEA, CAS and Hybrid Sugery. Patients will be given 100 mg of aspirin plus 75 mg of clopidogrel daily for at least 5 days before the hybird surgery procedure. If they had stenting procedure, they will receive a daily dose of 100 mg aspirin and 75 mg clopidogrel thereafter. If not, they will take either 100mg aspirin or 75mg clopidogrel daily for life.
  Groups: Hybrid Surgery

SUMMARY:
The short-term and long-term efficacy of recanalization therapy needs to be further confirmed by large-sample prospective studies. The comparison of success rate, complication rate and efficacy among the three recanalization modalities also needs to be further explored. The purpose of this cohort study is to observe the success rate, efficacy and safety of recanalization treatment for non-acute occlusion, and to further compare the advantages and disadvantages of CEA, endovascular intervention and hybrid surgery.

DETAILED DESCRIPTION:
Carotid artery occlusion is one of the primary causes of ischemic stroke. When the occlusion time exceeds 30 days, it is commonlly referred to as chronic carotid artery occlusion (CCAO), and patients with carotid artery occlusion over 24 hours are collectively referred as non-acute occlusion. Symptomatic non-acute occlusion patients with definite hemodynamic hypoperfusion still face a high risk of stroke recurrence under drug treatment, with recurrence rates reported to be between 12.3% and 22.7% within 2 years. Currently, the surgical methods for the treatment of carotid artery occlusion are mainly divided into extracranial-intracranial (EC-IC) bypass and recanalization treatment. Recanalization treatment includes CEA, endovascular intervention and hybrid surgery. While the Carotid Occlusion Surgery Study (COSS) and the recently published Carotid or Middle cerebral artery Occlusion Surgery Study (CMOSS) failed to reveal the significant advantages of EC-IC bypass surgery over medical treatment for patients with symptomatic artery occlusion combined with hemodynamic insufficiency, recanalization treatment has been shown to be a promising treatment modality by case-control studies with small sample size. However, the short-term and long-term efficacy of recanalization therapy needs to be further confirmed by large-sample prospective studies. The comparison of success rate, complication rate and efficacy among the three recanalization modalities also needs to be further explored. In addition, about half of non-acute occlusion patients have cognitive impairment, and the role of cerebral hemodynamics in cognitive impairment is still unclear. Therefore, the purpose of this cohort study is to observe the success rate, efficacy and safety of recanalization treatment for non-acute occlusion, and to further compare the advantages and disadvantages of CEA, endovascular intervention and hybrid surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Older than 18 years old;
2. Sign the informed consent form;
3. Carotid occlusion at least 24h;
4. Patients with clinical localization symptoms: ipsilateral hemisphere ischemia symptoms or ipsilateral eye ischemia symptoms or cognition impairment, with or without anterior circulation blood supply area infarction;
5. DSA confirmed common carotid artery or internal carotid artery (mTICI=0) occlusion;
6. Perfusion imaging confirms the presence of hypoperfusion in the corresponding area(CBF decrease);
7. The optimal medical treatment for patients who still have ischemic symptoms;
8. Routine DWI and ADC sequence examinations are performed before surgery no new infarction;

Exclusion Criteria:

1. Intracranial arteriovenous malformation or aneurysm;
2. Unstable angina, myocardial infarction (MI), or congestive heart failure in the last 6 months;
3. Uncontrolled diabetes mellitus defined as glucose > 300 mg/dL (16.67 mmol/L);
4. Patient is expected to have the ADP antagonist therapy interruption within 3 months after the procedure;
5. Pregnant or in the perinatal period;
6. Severe concomitant disease with poor prognosis (life expectancy < 3 years);
7. Intolerance or allergies to any of the study medications, such as aspirin or clopidogrel;
8. Allergy to iodine or radiographic contrast media;
9. Concomitant vascular conditions precluding endovascular;
10. Patients with large cerebral infarction within 2 weeks;
11. History of ipsilateral vocal cord paralysis;
12. Those with severe skin diseases who are expected to have difficulty healing the incision;
13. Poor functional status before onset (mRS score 4-5 points).
14. The area of infarction in the occluded vascular area exceeds half of the vascular supply area;
15. Already have dementia or psychiatric illness and are unable to complete neurological and cognitive assessments.
16. Any condition that in the surgeon's judgment suggests the patient an unsuitable surgical candidate.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People diagnosed with non-acute carotid occlusion, fulfilled the above eligible criteria in tertiary medical centers in China additionally will be enrolled consecutively.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-06-17 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Stroke or death whthin 30 days or recurrent ischemic stroke related of qualifying artery beyond 30 days through 12 months | Up to 12 months after procedure
  Including TIA, minor stroke, moderate stroke, severe stroke, and fatal stroke
MMSE within 30 and 90 days after procedure | 30 days and 90 days after procedure
  The Mini-Mental State Examination (MMSE) is a 30-point questionnaire that is used extensively in clinical and research settings to measure cognitive impairment. It is commonly used in medicine and allied health to screen for dementia. It is also used to estimate the severity and progression of cognitive impairment and to follow the course of cognitive changes in an individual over time; thus making it an effective way to document an individual's response to treatment. The MMSE's purpose has been not, on its own, to provide a diagnosis for any particular nosological entity.
MoCA scale within 30 and 90 days after procedure | 30 days and 90 days after procedure
  The Montreal Cognitive Assessment (MoCA) is a widely used screening assessment for detecting cognitive impairment.The MoCA test is a one-page 30-point test administered in approximately 10 minutes. The MoCA assesses: Short term memory/ Visuospatial abilities/ Executive functions/ Attention, concentration and working memory/ Language/ Orientation to time and place.

SECONDARY OUTCOMES:
Technical success rate | Up to 24 hours after procedure
  Defined as the target vessel residual stenosis less than 30% by CTA
Procedural success rate | Up to 24 hours after procedure
  Defines as the residual stenosis of the target vessel is less than 30% by CTA, and free of peri-procedural complications(includes cranial nerve injury, cardiac arrest, anaphylaxis, failure to recanalize blood vessels, distal embolism events, massive blood loss during operation, and residual thrombosis in the stent after operation)
Any stroke within 30 days, 90 days and 12 months after procedure | Within 30 days, 90 days and 12 months post-procedure
  Any stroke within 30 days, 90 days and 12 months
Death within 30 days, 90 days and 12 months after procedure | Within30 days, 90 days and 12 months post-procedure
  Death within 30 days, 90 days and 12 months
Cranial nerve injury | Within 30 days and 90 days post-procedure
  Number of participants who suffered from cranial nerve injury
Carotid artery or internal carotid artery reocclusion | Within 30 days, 90 days and 12 months post-procedure
  Number of participants who suffered from carotid artery or internal aryery rereocclusion (> 99%) detected by ultrasonography, CTA, MRA or DSA
Functional outcome | Within 30 days and 90 days post-procedure
  Functional outcome indicated by NIHSS (National Institutes of Health Stroke Scale: 0-42; 0 = no stroke 1-4 = minor stroke 5-15 = moderate stroke 15-20 moderate/severe stroke 21-42 = severe stroke ) or mRS (modified Rankin Scale: 0-6; 0-No symptoms at all. 1-No significant disability despite symptoms; able to carry out all usual duties and activities. 2-Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance. 3-Moderate disability; requiring some help, but able to walk without assistance. 4-Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance. 5-Severe disability; bedridden, incontinent and requiring constant nursing care and attention. 6-Dead.)
Other major complications | Within 30 days, 90 days and 12 months post-procedure
  Other major complications, such as myocardial infarction, pulmonary infection, postoperative bleeding, peri-procedural embolism, arterial dissection, vascular perforation, in-stent thrombus, post-procedural hyperperfusion syndrome, procedure related low perfusion infarction, etc.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Xuanwu Hospital, Capital Medical University., Beijing

IPD SHARING:
Plan to Share IPD: Undecided
Please contact the PI